CLINICAL TRIAL: NCT07399275
Title: Relationship Between Submental Tissue Oxygenation, Microvascular Reactivity, and Arterial Lactate During Major Surgical Procedures
Brief Title: Submental Tissue Oxygenation and Arterial Lactate in Major Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa Sevket Yilmaz Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gürcan Güler, Consultant Anesthesiologist and Intensivist, Bursa Sevket Yilmaz Training and Research Hospital
Other Study IDs: 2024-TBEK 2026/01-18
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Microcirculatory Dysfunction; Tissue Hypoperfusion; Microcirculatory Status; Microvascular Circulation; Near Infrared Spectroscopy; Vascular Occlusion Test; Lactate Blood Increase; Major Surgery
Keywords: tissue hypoperfusion; microvascular circulation; Near infrared spectroscopy; vascular occlusion; lactate blood increase; Major surgery
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major Surgery: Adult patients aged 18 years and older undergoing major surgical procedures under general anesthesia will be included in this cohort. Major surgery is defined as surgical procedures associated with a risk of significant blood loss and/or impaired tissue perfusion, requiring invasive arterial blood pressure monitoring and hourly arterial blood gas analysis. Eligible procedures include major abdominal, neurosurgical, and major orthopedic surgeries.
  All anesthetic and surgical management will be performed according to standard clinical practice. The study does not involve any experimental intervention or alteration of routine clinical care. Submental tissue oxygenation and microvascular reactivity will be monitored intraoperatively using non-invasive near-infrared spectroscopy techniques as part of observational data collection.
  Interventions: Other: No intervention. This is a prospective observational study. Near-infrared spectroscopy measurements are performed for monitoring purposes only and do not influence clinical management.

INTERVENTIONS:
Other: No intervention. This is a prospective observational study. Near-infrared spectroscopy measurements are performed for monitoring purposes only and do not influence clinical management. — This study does not include any therapeutic, diagnostic, or experimental intervention. It is a prospective observational study in which non-invasive near-infrared spectroscopy is used solely for intraoperative monitoring of submental tissue oxygenation and microvascular reactivity. Study measurements are collected for research purposes only and do not guide or alter anesthetic, surgical, or transfusion-related clinical decisions. All perioperative management is conducted according to standard institutional practice by the responsible clinical team.

SUMMARY:
During major surgical procedures performed under general anesthesia, changes in blood flow and oxygen delivery to tissues may occur due to blood loss, hemodynamic fluctuations, and anesthesia-related physiological effects. These changes can lead to impaired tissue perfusion, which is commonly reflected by increased arterial lactate levels. However, lactate measurements are intermittent and may not detect early perfusion abnormalities.

This prospective observational study aims to investigate the relationship between submental tissue oxygenation measured by near-infrared spectroscopy (NIRS), microvascular reactivity assessed by the vascular occlusion test, and arterial lactate levels during major surgery. Adult patients undergoing major abdominal, neurosurgical, or orthopedic procedures will be monitored intraoperatively using non-invasive NIRS techniques, while arterial blood gas analyses will be performed as part of routine clinical care.

The study does not involve any changes to standard anesthesia or surgical management. All treatments and clinical decisions will be made by the responsible care team according to routine practice. By evaluating non-invasive indicators of tissue oxygenation and microvascular function, this study aims to improve the understanding of early intraoperative tissue perfusion changes and their association with metabolic markers.

DETAILED DESCRIPTION:
This prospective, single-center, observational cohort study is designed to evaluate the relationship between intraoperative submental tissue oxygenation, microvascular reactivity, and arterial lactate levels during major surgical procedures performed under general anesthesia.

Major surgery is defined as procedures associated with a substantial risk of blood loss and/or tissue perfusion impairment, requiring invasive arterial blood pressure monitoring and hourly arterial blood gas analysis. Eligible surgical categories include major abdominal, neurosurgical, and major orthopedic procedures. Adult patients aged 18 years and older who meet the inclusion criteria will be enrolled.

All anesthetic and surgical management will be conducted according to standard clinical practice. The study protocol will not influence clinical decision-making. Hemodynamic management, fluid therapy, blood product transfusion, and ventilatory settings will be determined solely by the responsible anesthesia and surgical teams.

Intraoperative tissue oxygenation will be continuously monitored using near-infrared spectroscopy (NIRS). A NIRS sensor will be placed on the submental region, just inferior to the mandibular border and near the midline, after appropriate skin preparation. The sensor will be secured to minimize ambient light interference and motion artifacts. Baseline submental tissue oxygenation will be defined as the values obtained during a hemodynamically stable period of at least five minutes following anesthesia induction, without active surgical stimulation or significant fluctuations in mean arterial pressure.

Submental NIRS measurements will be recorded at 15-minute intervals throughout the intraoperative period, and hourly average and minimum values will be documented. A NIRS desaturation event will be defined as a decrease of 10% or more from baseline tissue oxygenation lasting for at least three minutes.

Microvascular reactivity will be assessed using the vascular occlusion test (VOT) applied to the thenar eminence of the non-dominant hand. A NIRS probe will be positioned on the thenar region following skin preparation. Transient arterial occlusion will be achieved using a non-invasive blood pressure cuff placed on the same upper extremity. The reoxygenation slope (ReO₂ slope) obtained during the reperfusion phase will be recorded as an indicator of microvascular reactivity. VOT measurements will be performed hourly during surgery and, whenever possible, synchronized with arterial blood gas sampling.

Arterial blood gas samples will be obtained hourly through an existing arterial catheter as part of routine intraoperative monitoring. Recorded parameters will include arterial lactate concentration, pH, base excess, hemoglobin, and hematocrit. Arterial lactate level will be considered the primary outcome measure of the study.

Intraoperative clinical data, including mean arterial pressure, vasopressor use, estimated blood loss, administered crystalloid and colloid fluids, and blood product transfusions, will be recorded on an hourly basis. For patients receiving blood transfusions, the indication for transfusion and timing of administration will be documented.

The intraoperative observation period will extend from anesthesia induction to the completion of surgery. All collected data will be analyzed to assess associations between submental tissue oxygenation, microvascular reactivity parameters, and arterial lactate levels over time. The study aims to explore whether non-invasive monitoring of tissue oxygenation and microvascular function may provide early insight into intraoperative tissue perfusion disturbances during major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Scheduled for major surgical procedures under general anesthesia
* Major surgery defined as procedures associated with a risk of significant blood loss and/or impaired tissue perfusion, requiring invasive arterial blood pressure monitoring and hourly arterial blood gas analysis
* Planned intraoperative arterial catheter placement as part of routine clinical care
* Ability to provide written informed consent

Exclusion Criteria:

* Age younger than 18 years
* Refusal or inability to provide informed consent
* Absence of invasive arterial blood pressure monitoring
* Known pregnancy
* Severe peripheral vascular disease affecting upper extremities
* Anatomical abnormalities or skin conditions preventing placement of NIRS sensors on the submental or thenar regions
* Emergency surgery requiring immediate intervention
* Preoperative severe metabolic acidosis (arterial pH < 7.20)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older undergoing major surgical procedures under general anesthesia at a single tertiary care center. Major surgery includes abdominal, neurosurgical, and major orthopedic procedures associated with a risk of significant blood loss and/or impaired tissue perfusion, requiring invasive arterial blood pressure monitoring and hourly arterial blood gas analysis as part of routine clinical care. All participants are enrolled prospectively and monitored intraoperatively without any alteration to standard anesthetic or surgical management.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between submental tissue oxygenation and arterial lactate levels | Intraoperatively, from anesthesia induction to the end of surgery
  The strength and direction of the association between intraoperative submental tissue oxygenation measured by near-infrared spectroscopy and arterial lactate levels during major surgery.

SECONDARY OUTCOMES:
Correlation between microvascular reactivity and arterial lactate levels | Intraoperatively, from anesthesia induction to the end of surgery
  The association between microvascular reactivity assessed by the vascular occlusion test (reoxygenation slope) and arterial lactate levels measured intraoperatively during major surgery.
Intraoperative submental NIRS desaturation events | Intraoperatively, from anesthesia induction to the end of surgery
  Occurrence of submental tissue oxygenation desaturation events, defined as a decrease of 10% or more from baseline lasting at least three minutes during the intraoperative period.
Relationship between submental tissue oxygenation and microvascular reactivity | Intraoperatively, from anesthesia induction to the end of surgery
  The association between intraoperative submental tissue oxygenation measured by near-infrared spectroscopy and microvascular reactivity assessed by the vascular occlusion test during major surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Principal Investigator — Department of Anesthesiology and Reanimation, Bursa Yuksek Ihtisas Training and Research Hospital, University of Health Sciences, Bursa
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker J, Nijsten MW, Jansen TC. Clinical use of lactate monitoring in critically ill patients. Ann Intensive Care. 2013 May 10;3(1):12. doi: 10.1186/2110-5820-3-12. PMID 23663301
- [Result] Gomez H, Mesquida J, Simon P, Kim HK, Puyana JC, Ince C, Pinsky MR. Characterization of tissue oxygen saturation and the vascular occlusion test: influence of measurement sites, probe sizes and deflation thresholds. Crit Care. 2009;13 Suppl 5(Suppl 5):S3. doi: 10.1186/cc8001. Epub 2009 Nov 30. PMID 19951387
- [Result] Scheeren TW, Schober P, Schwarte LA. Monitoring tissue oxygenation by near infrared spectroscopy (NIRS): background and current applications. J Clin Monit Comput. 2012 Aug;26(4):279-87. doi: 10.1007/s10877-012-9348-y. Epub 2012 Mar 31. PMID 22467064